CLINICAL TRIAL: NCT02776436
Title: Phase 1 Study to Evaluate the Safety of REducing the Prophylactic Dose of DEXamethasone Around Docetaxel Infusion in Patients With Early or Advanced Breast Cancer and Prostate Cancer
Brief Title: Reducing Dexamethasone Around Docetaxel Infusion
Acronym: REDEX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, J.R. Kroep, MD, PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: p15.157; 2015-000718-22 (EudraCT Number)
Record Dates: First submitted 2016-01-25; First posted 2016-05-18 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Dexamethasone; Absorptiometry, Photon; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast cancer (Experimental): Dose of prophylactic dexamethasone will be reduced as follows:
  STEP 1: 12 mg dexamethasone per day (8-4mg/day) for 3 days starting 1 day before administration. (n=6)
  STEP 2: 8mg dexamethasone per day (8mg once a day) for 3 days starting 1 day before administration. (n=6)
  STEP 3: day -1: 4 mg, day 0: 8 mg, day 1: 4 mg. (n=6)
  STEP 4: day -1: 0 mg, day 0: 8 mg, day 1: 4 mg. (n=6)
  STEP 5: day -1: 0 mg, day 0: 8 mg, day 1: 0 mg. (n=6)
  STEP 6: day -1: 0 mg, day 0: 4 mg, day 1: 0 mg. (n=6)
  Interventions: Drug: Dexamethasone
- Prostate cancer (Experimental): Dose of prophylactic dexamethasone will be reduced as follows:
  STEP 1: 2dd 8 mg at 12 and 1 hr before treatment (besides standard prednisone 5mg bid) (n=6)
  STEP 2: 8mg dexamethasone 1 hour before treatment (and standard prednisone 5mg bid). (n=6)
  STEP 3: 4mg dexamethasone 1 hour before treatment (and standard prednisone 5mg bid). (n=6)
  STEP 4: 0mg dexamethasone (only standard prednisone 5mg bid). (n=6)
  Interventions: Drug: Dexamethasone; Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone — Dose of prophylactic dexamethasone will be reduced for all patients
  Other Names: dexa
Drug: Prednisone — standard prednisone 5 mg bid for patients with prostate cancer
  Other Names: prednison
  Arms: Prostate cancer

SUMMARY:
The manufacturer recommends two different regimens of prophylactic dexamethasone to prevent hypersensitivity and fluid retention reactions caused by docetaxel: a 3-day regime of dexamethasone 8mg twice a day starting the day before chemotherapy for breast cancer and for prostate cancer 3 times 8mg dexamethasone on the day of docetaxel infusion, given the concurrent use of prednisone 2dd5mg. There is little evidence that supports this high dose regimen used nowadays. There is need to re-evaluate this high dosage of dexamethasone for three main reasons. First, dexamethasone can give side effects such as manifestation of latent diabetes mellitus, immunosuppression, personality changes, irritability, euphoria, or mania and mood swings. Second, dexamethasone is an immune suppressor, which might inhibit chemotherapy-induced apoptosis and compromise the efficacy of chemotherapeutic agents. Third, dexamethasone is a CYP3A4 inducer, which might increase docetaxel clearance. This study aims to evaluate the feasibility of reducing prophylactic of dexamethasone around docetaxel infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early breast cancer, or advanced breast cancer or prostate cancer patients receiving docetaxel (minimal 3 cycles monotherapy or in the regimen 4xAC > 4xdocetaxel or 3xFEC>3xdocetaxel or 6xTAC)
* Age ≥18 years
* WHO performance status 0-2
* Adequate bone marrow function: white blood cells (WBCs) ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function: bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL (<5 x UNL in case of liver metastases), Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥50 mL/min
* Survival expectation must be > 3 months
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Known hypersensitivity for docetaxel, paclitaxel or other chemotherapeutic agent or products containing polysorbate 80 or an earlier experience of anaphylaxis for food, insect bites, medication or another foreign substance.
* Existence of edema of the limbs or trunk or elsewhere localized.
* Active second malignancy
* Diabetes Mellitus
* Serious other diseases such as recent myocardial infarction (last 6 months), clinical signs of cardiac failure or clinically significant arrhythmias
* Female patients who are pregnant or breast-feeding
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Optimal dose/recommended dose (RD) of pre-medication dexamethasone around docetaxel infusion, dependent of occurrence of grade III/IV fluid retention and HSR according to the NCI CTCAE v4.03. | up to 30 weeks
  If one grade III/IV HSR or fluid retention reaction occurs in one of the six patients within one cohort, then three additional patients will be treated at that dose level. If there are no additional grade III/IV HSR or fluid retention in that additional 3 patients accrual to the next lower dose level will be started. If a grade III/IV HSR or fluid retention occurs in at least 2/6 or 2/9 patients, that dose will not be tolerated as safe and the last previous dose level of dexamethasone will be the RD.

SECONDARY OUTCOMES:
Glucose (mmol/L) response due to prophylactic dexamethasone on day 0 before chemotherapy. | up to 30 weeks
Insulin(mU/L), response due to prophylactic dexamethasone on day 0 before chemotherapy. | up to 30 weeks
IGF-1(nmol/L) response due to prophylactic dexamethasone on day 0 before chemotherapy. | up to 30 weeks
Number of participants with toxicity of chemotherapy according to NCI CTCAE v4.03 compared in each dose level of dexamethasone. | up to 30 weeks
Patient's quality of life (descriptive). | up to 30 weeks
Number of patients with single nucleotide polymorphisms in the glucocorticoid receptor. | one week

OTHER OUTCOMES:
The effect of dexamethasone on the Maximum concentration of docetaxel (Cmax) | 24 hours
The effect of dexamethasone on Area under the plasma-time concentration curve (AUC) of docetaxel. | 24 hours
The effect of dexamethasone on Elimination half-lives of docetaxel (T½,α; T½,β; T½,ƴ) of docetaxel. | 24 hours
The effect of dexamethasone on Total body clearance of docetaxel (Cl) of docetaxel. | 24 hours
The effect of dexamethasone on Volume of distribution of docetaxel at steady state (Vdss) | 24 hours

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Reinier de Graaf hospital, Delft
  - Leiden university medical center, Leiden
  - Haga hospital, The Hague

IPD SHARING:
Plan to Share IPD: No